CLINICAL TRIAL: NCT01132781
Title: The Effect of Theophylline in Patients With Allergic Rhinitis
Brief Title: Theophylline in Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2007ENT03; 2007-004642-32 (EudraCT Number)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Rhinosinusitis; Asthma; Allergic Rhinitis
Keywords: rhinosinusitis; asthma; allergic rhinitis; theophylline
MeSH Terms: conditions — Rhinosinusitis; Asthma; Rhinitis, Allergic | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 200mg twice daily of placebo drug
  Interventions: Drug: Placebo (Placebo Group)
- 200mg theophylline (Active Comparator): 200mg twice daily of slow release theophylline
  Interventions: Drug: Theophylline (Intervention Group)

INTERVENTIONS:
Drug: Theophylline (Intervention Group) — 200 mg twice daily of slow release theophylline
  Arms: 200mg theophylline
Drug: Placebo (Placebo Group) — 200 mg twice daily of placebo drug
  Arms: Placebo

SUMMARY:
Allergic rhinitis and asthma are common respiratory diseases, which often coexist. The prevalence of allergic rhinitis in subjects with asthma is up to 80%, and the prevalence of asthma is 3-5 times greater in subjects with rhinitis than healthy controls. The mechanisms of the allergen response in both diseases are parallel to each other, with similar mediator and cellular responses to similar allergens. These observations have led to the suggestion that both diseases are different expressions of one airway disease.We wish to evaluate the effect of low dose theophylline in patients with asthma, given its effects as subtherapeutic concentrations and the propensity to develop adverse events at higher doses.

DETAILED DESCRIPTION:
The disease modifying treatments for asthma and rhinitis mirror each other. The first line therapy being the topical corticosteroids, for which there is good evidence of superiority over other therapies. They work by altering the transcription of genes involved in the inflammatory process, thereby favourably influencing the synthesis of inflammatory proteins and cytokines. They have been shown to reduce the numbers of inflammatory cells and their inflammatory action. Other disease modifying therapies such as anti-IgE antibodies improve allergic symptoms in both asthma and rhinitis. Theophylline has been used for many years as a treatment for asthma but has not been used to help patients with rhinitis.

Theophylline has been considered a weak bronchodilator for many years. However relatively recently, it was shown to have anti-inflammatory effects in patients with asthma. It reduces eosinophil counts and eosinophilic cationic protein (ECP) concentration in induced sputum of asthmatic patients. The combination of low dose theophylline has greater effects on lung function and asthma severity than high dose inhaled corticosteroids.

Aubier el al have shown, using a nasal allergen challenge model of rhinitis, that 3 weeks treatment with slow release oral theophylline reduced the increase in the concentration of eosinophilic cationic protein (ECP) and the percentage of eosinophils in nasal lavage following the challenge. Furthermore there was a significant reduction in nasal symptoms in those patients treated with theophylline. However theophylline has not previously been evaluated as a therapeutic option in patients with chronic rhinitis in the clinic setting.

Cigarette smoking is a major cause of morbidity in patients with asthma and has been shown to be independently associated with impaired quality of life in asthmatic children. Recent evidence suggests that patients with asthma who smoke are relatively resistant to inhaled or oral corticosteroid therapy, with larger doses being required for clinical benefit. The actual mechanism for this observation is unknown however one hypothesis is that smoking has an effect on histone deacetylase. It is known that theophylline can active histone deacetylase and therefore improve the efficacy of corticosteroids.

Theophylline causes significant adverse effects at high doses. Unfortunately the bronchodilator effect occurs at doses very close to those causing adverse effects. This low therapeutic index for bronchodilation means that therapeutic monitoring is required. However the anti-inflammatory effect of theophylline and the effect of theophylline on histone deacetylase activity occurs at concentrations lower therapeutic level for bronchodilation.

Why have we chosen a dose of 200mg twice daily? In the study by Evans et al which compared low dose inhaled budesonide plus theophylline to high dose inhaled budesonide, greater effects with the theophylline combination were seen in terms of pulmonary function and hyperresponsiveness at serum concentrations of theophylline that were sub therapeutic (8.7mg/ml). Anti-inflammatory effects are seen in patients with chronic obstructive pulmonary disease at theophylline concentrations that are subtherapeutic. There have been studies in patients with asthma that have shown anti-inflammatory effects at in patients with asthma at doses of 250mg twice daily and 200mg twice daily. We wish therefore to evaluate the effect of low dose theophylline in patients with asthma, given its effects as subtherapeutic concentrations and the propensity to develop adverse events at higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged between 16 and 65 years.
* Weight between 50 and 150 Kg.
* Smokers, non-smokers or ex-smoker.
* Chronic rhinosinusitis as defined as 2 or more symptoms of nasal blockage/congestion, discharge, facial pain or reduction in smell for more than 12 weeks.
* A positive skin prick test or RAST to a perennial allergen
* Patients with a seasonal component to their symptoms can be enrolled out with the relevant pollen season.
* Patients must be receiving intranasal corticosteroids
* Patients will be permitted to receive inhaled short and long acting beta2 agonists or anti-cholinergic drugs, inhaled corticosteroids (up to a dose of 2mg per day BPD equivalent), oral montelukast or oral antihistamines.
* Able to provide written informed consent.

Exclusion Criteria:

* Significant medical, surgical or psychiatric disease that would affect the results of the study in the opinion of the investigator.
* Women who are pregnant or breast feeding
* Patients with previous cardiac problems or significant renal or hepatic impairment
* Upper respiratory tract infection in the last month as defined by yellow or green nasal discharge and increase in the usual nasal symptoms.
* Patients consuming more than the recommended amount of alcohol (14 units per week for women and 21 units per week for men) Inhaled corticosteroids at a dose greater than 2mg beclomethasone dipropionate (BDP) equivalent or oral corticosteroids or oral zafirlukast
* Currently receiving oral theophyllines.
* Previous adverse effects to oral or intravenous theophylline.
* Currently any medication known to interact with theophylline including

  * Allopurinol
  * Macrolide, quinolone or isoniazid
  * Fluvoxamine
  * Carbamazepine, phenytoin
  * Fluconazole or itraconazole
  * Barbiturates
  * Lithium
  * Oestrogens
  * Cimetidine

Ages: 16 Years to 65 Years | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Difference in total nasal symptom score | 18 weeks
  The primary endpoint will be the difference in total nasal symptom score between active and placebo treatment periods measured at the clinic

SECONDARY OUTCOMES:
The difference in domiciliary average total nasal symptom score | 18 weeks
The difference in nasal peak inspiratory flow at clinic visit | 18 weeks
  Nasal inspiratory flow will be measured using an In-check™ flow meter (Clement Clarke International Ltd, Harlow, UK). After blowing their nose, patients will inspire forcefully from residual volume to total lung capacity with their mouth closed. All measurements will be made while in the sitting position with a good seal around a purpose built facemask. The median of 3 readings will be recorded. For the purposes of the diary card data, these measurements will be recorded at 2200hrs. The average of the last 5 days measurements will be used in the analysis.
The difference in domiciliary nasal peak inspiratory flow | 18 weeks
  Nasal inspiratory flow will be measured using an In-check™ flow meter (Clement Clarke International Ltd, Harlow, UK). After blowing their nose, patients will inspire forcefully from residual volume to total lung capacity with their mouth closed. All measurements will be made while in the sitting position with a good seal around a purpose built facemask. The median of 3 readings will be recorded. For the purposes of the diary card data, these measurements will be recorded at 2200hrs. The average of the last 5 days measurements will be used in the analysis.
The difference in Sino-Nasal Outcomes Test (SNOT) -22 questionnaire | 18 weeks
  The Sino-Nasal Outcomes Test (SNOT) is a validated disease-specific health-related quality of life instrument. It comprises 22 questions and takes less than 5 minute to complete. It is self administered questionnaire. It will be completed at each study visit.
Secondary Analysis | 18 weeks
  A secondary analysis will be undertaken to determine whether there is a difference in primary and secondary endpoints (above) between treatment with theophylline and placebo in patients who smoke versus those who do not smoke.
Serum theophylline concentration at the end of both placebo or active treatment periods. | 18 weeks
Serum urea and electrolyte concentration at the both placebo or active treatment periods | 18 weeks
Drug related adverse effects | 18 weeks
The difference histone deacetylase activity from epithelial cells obtained from nasal scrapings. | 18 weeks
  Nasal scrapings will be taken from the right nostril using a Rhino-probe Nasal Mucosal Curette (Arlington Scientific Inc, Springville, Utah, USA). Two scrapes will be taken under direct vision according to manufacturer's guidelines. These will be taken at visits 3 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom